CLINICAL TRIAL: NCT04408339
Title: COVID-19 Disease in Cancer Patients: Evaluation of Clinical Course and Impact on Oncological Care in the Hamburg Metropolitan Area Including Prospective Biobanking
Brief Title: COVID-19 in Cancer Patients: Evaluation of Clinical Course and Impact on Oncological Care Including Biobanking
Acronym: COVIDHELP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hopsital Schleswig Holstein Campus Lübeck (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Other Study IDs: PV7313
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cancer; COVID
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The COVIDHELP study will prospectively evaluate the yet unknown clinical course of the COVID-19 infection in cancer patients and document the impact of potential infrastructural limitations on cancer care of COVID-19 positive patients. All patients consenting will provide peripheral blood samples for prospective biobanking with the aim of investigating immune response and immunity against COVID-19.

DETAILED DESCRIPTION:
Based on patients, who are treated in the University Cancer Center Hamburg (UCCH) and its contracted partner network, which comprises all cancer treating departments at the University Medical Center of Hamburg-Eppendorf (UKE), as well as 19 office-based oncologists and 20 surrounding hospitals, recruitment for the study will be done as follows:

(i) as a cancer patient during regular aftercare appointments who reports a current or past COVID-19 infection.

(ii) as an acute COVID-19 patient who reports a prevalent cancer diagnosis

Data will be collected as available from routine clinical care and includes demographic and biometric data, medical history, baseline data at inclusion as well as inpatient and intensive care unit admissions. Upon consent, patients will provide peripheral blood samples at time of inclusion and after 6 month. Recruitment is limited to a one-year period (April 2020 - April 2021).

ELIGIBILITY:
Key inclusion criteria:

* Known diagnosis of cancer
* Known diagnosis of CoVID-19 infection
* Age ≥ 18 years
* Signed informed consent

Key exclusion criteria:

• refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population consists of patients, who are treated in the University Cancer Center Hamburg (UCCH) and its contracted partner network, who are either cancer patients reporting a current or past COVID-19 infection, or acute COVID-19 patients who report a prevalent cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-14 (Estimated); Study Completion 2022-04-14 (Estimated)

PRIMARY OUTCOMES:
Rate of hospitalization | 2 years
  Measured in percentage
Duration of hospitalization | 2 years
  Measured in days from date of admission to definitive discharge
Rate of admission to intensive care unit | 2 years
  Measured in percentage
Length of stay in intensive care unit | 2 years
  Measured in days from date of admission to intensive care unit to the date of discharge
Need of mechanical ventilation | 2 years
  Measured in percentage
Duration of mechanical ventilation | 2 years
  Measured in days from the date of intubation to the stop date of mechanical ventilation
Disease-specific mortality rate | 2 years
  COVID-19 associated mortality rate

SECONDARY OUTCOMES:
Rate of patients, whose oncologic treatment had to be modified due to COVID-19 | 2 years
  Measured in percentage. Modification is defined as cancellation, postponement or dose-adjustment of treatment.
Cellular and humoral immune response to COVID-19 infection | 6 month
  Analysis of blood samples at time of diagnosis and after 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Katja Weisel, MD, Principal Investigator — University Medical Center of Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data will be shared